CLINICAL TRIAL: NCT06991439
Title: A Qualitative Study on the Experiences of Mental Healthcare Workers Using STAPP@Work: A Mobile Self-Management Application to Support Work-Related Stress
Brief Title: Qualitative Exploration of a Mobile Stress Management Intervention for Mental Health Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevda Demirel (Other)
Collaborators: GGZ Centraal (Other)
Responsible Party: Sponsor-Investigator, Sevda Demirel, PhD Candidate, GGZ Centraal
Organization: GGZ Centraal (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S@W_240101
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Work-Related Stress; Coping Behaviour; User Experience of Mobile Application
Keywords: User Experiences; Work-related stress; Self-management; Stress management; Mobile Health; mHealth; Qualitative study; Self-Monitoring; Mental Healthcare Workers; Healthcare Professionals
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: All participants are assigned to use the STAPP@Work mobile intervention for a two-week period. There is no comparison or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAPP@Work App Intervention (Experimental): Participants assigned to this arm will use the STAPP@Work mobile intervention for a period of two weeks. The app prompts users multiple times per day to self-monitor their stress by answering short questions about their current activity, mood, and stress signals. It provides real-time feedback, visual summaries of stress patterns over time, and practical tips for stress management. After the intervention period, participants will take part in a semi-structured interview to reflect on their experiences of using the app.
  Interventions: Device: A self-monitoring mobile application for stress management at work

INTERVENTIONS:
Device: A self-monitoring mobile application for stress management at work — STAPP@Work is a digital self-monitoring intervention designed for the workplace to manage work-related stress. The app prompts users multiple times per day to self-monitor their stress by answering short questions about their current activity, mood, and stress signals. It provides real-time feedback, visual summaries of stress patterns over time, and practical tips for stress management.

SUMMARY:
The goal of this qualitative intervention study is to explore the experiences of mental healthcare workers using the STAPP@Work app to manage work-related stress. STAPP@Work is a mobile self-monitoring app designed for the workplace, that supports users in recognizing, understanding, and managing daily stress. The app measures stress levels multiple times per day by asking what you were doing, how you were feeling and your stress signals. It offers real-time feedback and a visual overview of stress levels at both the daily and weekly level, including the context. This allows users to recognize their own stress triggers and patterns. In addition, the app provides practical suggestions to help users cope with stress.

The main question this study aims to answer is:

- How do mental healthcare workers experience the use of the STAPP@Work app in daily work life?

Participants will:

* Use the STAPP@Work app for a period of 2 weeks.
* Participate in a semi-structured interview after the use of the intervention to discuss their experiences with the app.

This is a single-group qualitative study. There is no control or comparison group. The findings will contribute to understanding how mobile health interventions can support employees in high-pressure healthcare environments, and provide insight into user experiences, perceived benefits and limitations, and factors that may influence engagement and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Employee at GGz Centraal

Exclusion Criteria:

* Not employed at GGz Centraal
* Prior participation in a STAPP@Work research study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Perceived Impact of the STAPP@Work App on Stress Recognition | Shortly after completion of the 2-week intervention (target: within 1 week)
  Assessed through qualitative analysis of post-intervention interviews focusing on participants' experiences of using the STAPP@Work app during work.
Perceived Impact of the STAPP@Work App on Coping Behaviour | Shortly after completion of the 2-week intervention (target: within 1 week)
  Assessed through qualitative analysis of post-intervention interviews focusing on participants' experiences of using the STAPP@Work app during work.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Roke, MD, PhD, Principal Investigator — GGZ Centraal
Locations (1):
- GGZ Centraal, Almere Stad, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no public individual participant data sharing is planned, but data may be made available upon reasonable request from the corresponding author, in accordance with institutional and ethical guidelines.

REFERENCES:
- [Background] Demirel S, Roke Y, Hoogendoorn AW, Hoefakker J, Hoeberichts K, van Harten PN. Assessing the Effectiveness of STAPP@Work, a Self-Management Mobile App, in Reducing Work Stress and Preventing Burnout: Single-Case Experimental Design Study. J Med Internet Res. 2024 Feb 29;26:e48883. doi: 10.2196/48883. PMID 38275128